CLINICAL TRIAL: NCT05358951
Title: Sleep Treatment Education Program for Young Adult Cancer Survivors (STEP-YA): An Online Educational Intervention for Insomnia
Brief Title: Sleep Treatment Education Program for Young Adult Cancer Survivors (STEP-YA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Recklitis, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-613; R21CA261863 (NIH)
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Insomnia; Insomnia Due to Medical Condition; Cancer
Keywords: Insomnia; Insomnia Due to Medical Condition; Cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NON-COACHING CONDITION STEP-YA (Active Comparator): Participants will receive a single online education session and complete online questionnaires then be randomized to not receive additional coaching support sessions.
  Participates will also complete follow up questionaires at 4 and 8 weeks post baseline.
  Interventions: Behavioral: STEP-YA without Coaching
- COACHING CONDITION STEP-YA (Experimental): Participants will receive a single online education session and complete online questionnaire then be randomized to receive 2 individualized remote coaching sessions.
  Participates will also complete follow up questionaires at 4 and 8 weeks post baseline.
  Interventions: Behavioral: STEP-YA with Coaching

INTERVENTIONS:
Behavioral: STEP-YA with Coaching — Online instruction on behavioral changes to improve sleep with 2 additional individually coached session
  Arms: COACHING CONDITION STEP-YA
Behavioral: STEP-YA without Coaching — Online instruction on behavioral changes to improve sleep without additional individually coached session
  Arms: NON-COACHING CONDITION STEP-YA

SUMMARY:
The purpose of the study is to learn if a single online education session, with or without individualized coaching sessions, can help improve young adult cancer survivors' (YACS) sleep.

The name of the study intervention is Sleep Treatment Education Program for Young Adult Cancer Survivors (STEP-YA).

DETAILED DESCRIPTION:
This study is a randomized controlled trial of young adult cancer survivors with clinically significant symptoms of insomnia to evaluate the cognitive-behavioral based Sleep Treatment Education Program for Young Adult Cancer Survivors (STEP-YA).

All participants will take part in a single STEP-YA session, during which they will complete baseline measures prior to randomization and then receive the STEP-YA intervention. Participants will then be randomly assigned to receive the STEP-YA intervention either, 1) alone (non-coaching condition), or 2) with the addition of 2 remote coaching sessions (coaching condition). Participants will also complete follow-up measures 4 and 8 weeks post-baseline.

It expected that about 74 people will take part in this study

ELIGIBILITY:
Inclusion Criteria:

To be determined by patient self-report from eligibility screening with potential participants. (See Appendix A for eligibility screening materials). Participants must be screened for eligibility ≤2 weeks prior to study enrollment. Participants who are screened earlier must be rescreened within this period.

* Age 20-39
* History of a cancer diagnosis (except non-melanoma skin cancer) ≥ 1 year prior
* No active cancer therapy (excluding chemoprevention) in the past four months, and no further therapy planned
* Significant insomnia as evidenced by an Insomnia Severity Index score ≥12
* Able to read and write in English

Exclusion Criteria:

* Survivors who report ever being diagnosed with Bipolar Disorder.
* Survivors who report ever being diagnosed with a Seizure Disorder or have experienced a seizure in the past 12 months.
* Intention to adjust (decrease or increase) use of any prescribed or over-the-counter medications taken to decrease insomnia during the study period.
* Survivors who report being diagnosed with sleep apnea who are not receiving recommended medical treatment for their sleep apnea (as assessed by screening questions, see Appendix A).
* Survivors who report suspected sleep apnea who have not completed an evaluation by a sleep specialist (as assessed by screening questions, see Appendix A).
* Survivors who report their usual bedtime does not fall between 5:00 pm and 5:00 am.
* Employment that involves irregular sleep patterns, such as shift-work or frequent long-distance travel across time zones, or employment in a position that could impact public safety (such as air traffic-controller, operating heavy machinery)
* Any impairment (e.g., hearing, visual, cognitive) that interferes with the ability to complete all study procedures independently.
* Prior participation in a research study which provided an educational or behavioral intervention for insomnia
* Prior participation in a behavioral treatment or patient education program for insomnia delivered at the Dana-Farber Cancer Institute, or at Boston Children's Hospital.
* Participation in behavioral or educational interventions for insomnia in the 2 years prior to enrollment. This includes in-person as well as synchronous and asynchronous online insomnia programs, but not independent use of books, workbooks or other written self-help materials addressing insomnia.

Ages: 20 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2022-11-19 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Change at 8 Weeks | Baseline to 8-weeks post-intervention session
  The Insomnia Severity Index (ISI), a 7-item self-report questionnaire assessing severity, and impact of insomnia symptoms will be used.

SECONDARY OUTCOMES:
Profile of Mood States Change at 8 weeks | Baseline to 8-weeks post-intervention session
  The Profile of Mood States - Short Form (POMS-SF), a 35-item measure of participant mood states that provides multiple scales including an overall Total Mood Disturbance (TMD) score will be used
Profile of Mood States Change at 4 weeks | Baseline to 4-weeks post-intervention session
  The Profile of Mood States - Short Form (POMS-SF), a 35-item measure of participant mood states that provides multiple scales including an overall Total Mood Disturbance (TMD) score will be used
Insomnia Severity Change at 4 weeks | Baseline to 4-weeks post-intervention session
  The Insomnia Severity Index (ISI), a 7-item self-report questionnaire assessing severity, and impact of insomnia symptoms will be used.

OTHER OUTCOMES:
Insomnia Severity at 16 weeks (optional) | 16 weeks post-intervention session
  The Insomnia Severity Index (ISI), a 7-item self-report questionnaire assessing severity, and impact of insomnia symptoms will be used.
Initial Satisfaction with Intervention Session | Up to 4 weeks post-intervention
  Study specific questionnaire assessing intervention acceptability, credibility and participant satisfaction
Satisfaction with Coaching Sessions | Up to 4 weeks post-intervention
  Study specific questionnaire describing satisfaction with coaching sessions
Final satisfaction with the intervention | 8 Weeks post-intervention session
  Study specific questionnaire asking about participant satisfaction with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Recklitis, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Michaud AL, Bice B, Miklos E, McCormick K, Medeiros-Nancarrow C, Zhou ES, Recklitis CJ. Sleep Treatment Education Program for Young Adult Cancer Survivors (STEP-YA): Protocol for an Efficacy Trial. JMIR Res Protoc. 2023 Nov 29;12:e52315. doi: 10.2196/52315. PMID 38019571